CLINICAL TRIAL: NCT04041492
Title: Effect of Supplementation With Vitamins D3 and K2 in Non-carboxyled Osteocalcine and Insulin Serum Levels in Patients With Diabetes Mellitus Type 2
Brief Title: Effect of Vitamins D3 and K2 in uOc and Insulin Serum Levels in Patients With Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Julio Ivan Aguayo Ruiz, Principal Investigator, University of Guadalajara
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Supportive Care
Other Study IDs: F-2017-1702-14
Record Dates: First submitted 2019-07-31; First posted 2019-08-01 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Diabetes Mellitus, Type 2; Bone Loss; Insulin Resistance
Keywords: diabetes; osteocalcin; insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Bone Diseases, Metabolic; Insulin Resistance; Diabetes Mellitus | interventions — Dietary Supplements

STUDY DESIGN:
Intervention Model Description: Controlled clinical trial, with randomization simple, double blind.
Who Masked: Participant, Care Provider, Investigator
Masking Description: randomization simple, double blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Vitamin D3 1000UI + Placebo (Calcined Magnesia).
  Interventions: Dietary Supplement: Supplementation with Vitamin D3 y K2
- Group 2 (Experimental): Vitamin K2 100 mcg + Placebo (Calcined Magnesia).
  Interventions: Dietary Supplement: Supplementation with Vitamin D3 y K2
- Group 3 (Active Comparator): Vitamin D3 1000UI + Vitamin K2 100 mcg
  Interventions: Dietary Supplement: Supplementation with Vitamin D3 y K2

INTERVENTIONS:
Dietary Supplement: Supplementation with Vitamin D3 y K2 — Supplementation at a dose of 1 capsule every 24 hours x 3 months

SUMMARY:
Introduction: Patients with DM2 have chronic hyperglycemia derived from a decrease in insulin sensitivity, cause of comorbidities such as bone demineralization, decreasing quality of life and increasing mortality. This could be related to changes in the serum levels of carboxylated Osteocalcin and Insulin, together with the deficit the daily consumption of vitamins D3 and K, which is crucial for the process of mineralization of the bone matrix.

Research question: What is the effect of supplementation with Vitamins D3 and K2 on serum levels of Carboxylated Osteocalcin and Insulin in patients with Type 2 Diabetes mellitus?

Hypothesis: Supplementation with Vitamins D3 and K2 modifies the serum levels of Carboxylated Osteocalcin and Insulin in patients with Type 2 Diabetes mellitus.

General Objectives: To assess the effect of supplementation with Vitamins D3 and K2 on serum levels of Carboxylated and Non-Carboxylated Osteocalcin in patients with Type 2 Diabetes mellitus.

Material and Methods: Clinical trial, double blind, randomization, 40 patients with DM2, 35-65 years, supplementation (3 months), clinical and laboratory determinations (uOC and Insulin).

* Group 1: Vitamin D3 1000UI + Placebo
* Group 2: Vitamin K2 100 mcg + Placebo
* Group 3 (Positive Control): Vitamins D3 1000UI + K2 100 mcg

DETAILED DESCRIPTION:
Type 2 diabetes mellitus is a group of metabolic disorders characterized by chronic hyperglycemia, being one of the main causes of mortality in our country.

There are different comorbidities, including bone demineralization, which involve an imbalance in the process of bone formation and resorption, which entails the risk of decreasing bone mineral density. These processes could be related to the serum levels of Non-carboxylated Osteocalcin and Insulin, said molecule locally modulates the process of bone mineralization.

On the other hand, it is known that the daily consumption of vitamins in a general diet in our population (specifically including vitamins D3 and K), is below the necessary basic requirements, so considering crucial elements for the benefit of Bone matrix mineralization, which is why the present study proposes supplementation with the aforementioned vitamins in patients with Type 2 DM, to avoid a decrease in bone mineral density, increasing the mortality rate of individuals suffering from it.

1. - The study subjects from the West of the country were invited to participate in the research protocol, where their objective was explained and the signing of the consent was requested under information, where a structured evaluation was subsequently carried out consisting of :

   a) Comprehensive clinical evaluation (including general sociodemographic data of a complete medical history).
2. - Once the previous data was obtained, the randomization of the treatment was carried out, classifying the patients in the following groups:

   * Group 1 Vitamin D3 1000UI + Placebo (Calcined Magnesia).
   * Group 2 Vitamin K2 100 mcg + Placebo (Calcined Magnesia).
   * Group 3 (Positive Control) Vitamins D3 1000UI + K2 100 mcg.
3. - Blood sample collection through Punzocat, which was placed in a red tube, for subsequent centrifugation at 3500rpm x 15 minutes, performing aliquots of the serum obtained and stored at -80 ° C and thus perform the pertinent quantifications of the molecules to study.
4. - Quantification of serum levels of non-carboxylated Osteocalcin and Insulin

   a) The determinations corresponding to the serum levels of Non-carboxylated Osteocalcin and Insulin were made, both baseline prior to the intervention as well as the final quantification, once the supplementation was finished, by means of the indirect ELISA technique (commercial reagents -Takara were used - for the realization of these determinations), which involved the following process: In a plate the wells were coated with a first antibody, then a wash was performed to remove the excess antibody, after that, the sample in which the antigen was found was added, which was retained in the well after being recognized by the first antibody, a second wash was subsequently made to remove unbound material, then a solution with a second labeled anti-antigen antibody was applied. Thus each antigen molecule was bound to an antibody in the base that kept it fixed and a second antibody for its reaction and labeling. Finally, the plate was introduced into a spectophotometer and the absorbance was measured at a length of 450 nm, for both non-carboxylated Osteocalcin and Insulin.
5. - The quantification in serum of cholesterol and triglycerides was carried out by using the fully automated random access analyzer equipment for clinical chemistry, model ERBA XL 200.
6. - The evaluation of the HOMA index was calculated by using the equations HOMA-IR and HOMA-B, for insulin resistance (IR) and Percentage, respectively.
7. - The daily of adherence to treatment was provided, so that they recorded all those important events that would ensure adequate intake of vitamins, as well as adverse reactions to them, which were evaluated in scheduled appointments, in addition to each The corresponding bottles were delivered consecutively for each of the 3 months of intervention, with the corresponding vitamins for each patient according to their allocation group.
8. - Finally, in the last visit the results obtained during the whole study were made known to each of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Originating and residents of Western Mexico
* Both genres
* Age of 30-75 years
* Diagnosis of DM2 (ADA Criteria) of at least 5 years of evolution
* Sign an informed consent letter.

Exclusion Criteria:

* Use of active drugs for bone mineralization
* Pregnancy
* Lactation
* Creatinine or transaminase more than double the upper limit
* Diet added with calcium or vitamins (D, K).

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2018-02-14 (Actual); Study Completion 2019-02-14 (Actual)

PRIMARY OUTCOMES:
Non-carboxylated osteocalcin | 3 months
  Serum levels
Insulin | 3 months
  Serum levels

SECONDARY OUTCOMES:
Weight | 3 months
  kg
Height | 3 months
  m
Body mass index | 3 months
  Quetelet index
HOMA Index | 3 months
  Insulin resistance

CONTACTS AND LOCATIONS:
Locations (1):
- Julio Iván Aguayo, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No
Non-sharable data

REFERENCES:
- [Derived] Aguayo-Ruiz JI, Garcia-Cobian TA, Pascoe-Gonzalez S, Sanchez-Enriquez S, Llamas-Covarrubias IM, Garcia-Iglesias T, Lopez-Quintero A, Llamas-Covarrubias MA, Trujillo-Quiroz J, Rivera-Leon EA. Effect of supplementation with vitamins D3 and K2 on undercarboxylated osteocalcin and insulin serum levels in patients with type 2 diabetes mellitus: a randomized, double-blind, clinical trial. Diabetol Metab Syndr. 2020 Aug 18;12:73. doi: 10.1186/s13098-020-00580-w. eCollection 2020. PMID 32831908